CLINICAL TRIAL: NCT00199563
Title: The Use and Efficacy of Sildenafil in Diabetic Men With Erectile Dysfunction: the Impact on Endothelial Function, a Pilot Feasibility Study
Brief Title: Use of Sildenafil (Viagra) in Diabetic Men With Erectile Dysfunction: the Impact on Blood Vessels
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: R-04-402; Ethics Review: 10331; R-04-402 (Other: Lawson Research Institute)
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Impotence
Keywords: Viagra; sildenafil
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- active drug (Active Comparator): Viagra 100 mg / daily for 12 weeks.
  Interventions: Drug: Viagra
- Placebo (Placebo Comparator): placebo/daily for 12 weeks
  Interventions: Drug: Viagra

INTERVENTIONS:
Drug: Viagra — Sildenafil 100mg daily for 12 weeks
  Other Names: Sildenafil

SUMMARY:
* To evaluate the impact of nightly sildenafil vs placebo use on diabetic men with and without proven endothelial dysfunction and coexisting erectile concerns.
* To determine if chronic sildenafil use compared to placebo positively impacts endothelial function among a cohort of diabetic mend with erectile dysfunction
* To assess the salvage rate of sildenafil - failures who demonstrate improved response rates over time with chronic use
* To assess if microalbuminuria predicts flow-mediated dilation (FMD) response
* To measure and identify if other patient specific characteristics predict for sildenafil erectile response and flow-mediated dilatation (FMD) response over time (patient specifics; blood pressure, HBA1c, weight, BMI, age IIEF score at baseline)

DETAILED DESCRIPTION:
60 type II diabetic men with erectile dysfunction will be enrolled in this trial, evaluated over a 12 week period. Randomization into one of two arms (placebo, daily sildenafil 50mg) will be a doubly blinded. Subjects will be followed by IIEF, diaries and brachial forearm medial dilatation duplex scans, urinary microalbuminuria and serum chemistry.

Study time-points are at baseline, 6 and 12 weeks.

Study participants will be instructed to use the study medication at the specified frequency but will be allowed flexibility to suit their erectile needs.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Type 2 diabetes > 6 months in duration. Men using oral hypoglycemic agents and /or insulin will be permitted into the trial.
* Stable hetero- sexual relationship for > 6 months
* IIEF score at baseline <21·
* Agrees to sign informed consent

Exclusion Criteria:

* Known hypersensitivity to sildenafil
* Use of nitrates
* Use of anti-coagulants
* History of significant heart disease, +/or myocardial infarction within last 6 months
* Unable to understand or unwilling to sign informed consent
* Concomitant use of erectogenic agent during study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2004-08; Primary Completion 2007-10 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Determine if PDE5 use over 12 week period in ED diabetic men improves endothelial function as measured by FMD of the brachial artery, as compared to placebo; Assess treatment response to sildenafil over a 12 week period of exposure compared to placebo. | 12 weeks

SECONDARY OUTCOMES:
IIEF Questionnaire & diary response;Blood pressure and microalbuminuria; Side effects | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerald B Brock, MD, Principal Investigator — Lawson Health Research Institute/St. Joseph's Health Care London
Locations (1):
- St. Joseph's Health Care London/Urology Clinic, London, Ontario, Canada

REFERENCES:
- [Result] Yu HI, Sheu WH, Lai CJ, Lee WJ, Chen YT. Endothelial dysfunction in type 2 diabetes mellitus subjects with peripheral artery disease. Int J Cardiol. 2001 Mar;78(1):19-25. doi: 10.1016/s0167-5273(00)00423-x. PMID 11259809
- [Result] De Angelis L, Marfella MA, Siniscalchi M, Marino L, Nappo F, Giugliano F, De Lucia D, Giugliano D. Erectile and endothelial dysfunction in Type II diabetes: a possible link. Diabetologia. 2001 Sep;44(9):1155-60. doi: 10.1007/s001250100616. PMID 11596671
- [Result] Feldt-Rasmussen B. Microalbuminuria, endothelial dysfunction and cardiovascular risk. Diabetes Metab. 2000 Jul;26 Suppl 4:64-6. PMID 10922975
- [Result] Desouza C, Parulkar A, Lumpkin D, Akers D, Fonseca VA. Acute and prolonged effects of sildenafil on brachial artery flow-mediated dilatation in type 2 diabetes. Diabetes Care. 2002 Aug;25(8):1336-9. doi: 10.2337/diacare.25.8.1336. PMID 12145231
- [Result] Dishy V, Sofowora G, Harris PA, Kandcer M, Zhan F, Wood AJ, Stein CM. The effect of sildenafil on nitric oxide-mediated vasodilation in healthy men. Clin Pharmacol Ther. 2001 Sep;70(3):270-9. doi: 10.1067/mcp.2001.117995. PMID 11557915
- [Result] Katz SD, Balidemaj K, Homma S, Wu H, Wang J, Maybaum S. Acute type 5 phosphodiesterase inhibition with sildenafil enhances flow-mediated vasodilation in patients with chronic heart failure. J Am Coll Cardiol. 2000 Sep;36(3):845-51. doi: 10.1016/s0735-1097(00)00790-7. PMID 10987609